CLINICAL TRIAL: NCT02525653
Title: A Phase II Trial of Albumin-Bound Paclitaxel and Gemcitabine in Patients With Untreated Stage IV or Recurrent Squamous Cell Lung Cancers
Brief Title: Albumin-Bound Paclitaxel and Gemcitabine in Patients With Untreated Stage IV or Recurrent Squamous Cell Lung Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Celgene Corporation (Industry); Miami Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-054
Record Dates: First submitted 2015-08-14; First posted 2015-08-17 (Estimated); Results first posted 2020-05-08 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2019-09

CONDITIONS: Lung Cancer; Untreated Stage IV or Recurrent Squamous Cell Lung Cancers
Keywords: Albumin-Bound; Paclitaxel; Gemcitabine; 15-054
MeSH Terms: conditions — Lung Neoplasms | interventions — Albumin-Bound Paclitaxel; Gemcitabine

ARMS (1):
- Albumin-Bound Paclitaxel and Gemcitabine (Experimental): During each 21-day cycle, albumin-bound paclitaxel at 100mg/mg2 over 120 minutes and gemcitabine at 1000mg/m2 over 30 minutes will be given intravenously on days 1 and 8 of each 21 day cycle. Treatment will continue until disease progression or intolerable side effects. After the 4th cycle of treatment, patients will have the option of discontinuing gemcitabine and proceeding with weekly albumin-bound paclitaxel as maintenance therapy.
  Interventions: Drug: albumin-bound paclitaxel; Drug: gemcitabine

INTERVENTIONS:
Drug: albumin-bound paclitaxel
Drug: gemcitabine

SUMMARY:
The purpose of this study is to test the safety and effectiveness of albumin-bound paclitaxel plus gemcitabine in patients with advanced squamous cell lung cancers. The investigators would like to determine the percentage of patients with squamous cell lung cancers who experience shrinkage of their tumors following treatment with this regimen. This combination of drugs is not a standard therapy for patients with squamous cell lung cancers. However, each of these drugs, when given alone or with other chemotherapies, is FDA-approved for the treatment of this disease.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell lung cancer
* Newly diagnosed untreated Stage IV and/or recurrent after adjuvant therapy with metastatic disease
* Patients previously treated with immune checkpoint inhibitor therapy are eligible
* Measurable disease as per RECIST 1.1
* Greater than 6 months since receiving neo-adjuvant or adjuvant chemotherapy.
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Women of childbearing potential and sexually active men enrolled in the study must agree to practice effective contraception method during treatment and for three months after completing treatment
* Negative serum or urine β-hCG pregnancy test at screening for patients of childbearing potential
* < Grade 2 pre-existing peripheral neuropathy (per CTCAE)
* Marrow and organ function as follows:
* ANC ≥ 1500 cells/mm3
* Platelets > 100,000 cells/mm3
* Hemoglobin>9g/dL
* Creatinine clearance ≥ 40mL/min
* Bilirubin ≤ 1.5 mg/dL
* AST/ALT≤2.5 x upper limit of normal range (ULN),
* alkaline phosphatase ≤ 2.5 X upper limit of normal, unless bone metastasis in present in the absence of liver metastasis

Exclusion Criteria:

* Prior treatment with albumin-bound paclitaxel or gemcitabine
* Prior systemic anticancer therapy for advanced squamous cell lung cancer
* Untreated brain metastasis. Patients with treated brain metastases who are off steroids are eligible
* Peripheral neuropathy greater than grade 1
* Malignancies within the past 5 years other than non-melanoma skin cancer or insitu cervical cancer status post treatment
* Patients with other serious medical illnesses including, ongoing or active infection, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements
* Class III or IV congestive heart failure by New York Heart Association

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Paik, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Miami Cancer Institute Baptist Health South Florida, Miami, Florida
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York
  - Memorial Sloan Kettering Westchester, Sleepy Hollow, New York

REFERENCES:
- [Derived] Paik PK, Kim RK, Ahn L, Plodkowski AJ, Ni A, Donoghue MTA, Jonsson P, Villalona-Calero M, Ng K, McFarland D, Fiore JJ, Iqbal A, Eng J, Kris MG, Rudin CM. A Phase II Trial of Albumin-Bound Paclitaxel and Gemcitabine in Patients with Newly Diagnosed Stage IV Squamous Cell Lung Cancers. Clin Cancer Res. 2020 Apr 15;26(8):1796-1802. doi: 10.1158/1078-0432.CCR-19-3060. Epub 2020 Jan 9. PMID 31919132
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Albumin-Bound Paclitaxel and Gemcitabine
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Albumin-Bound Paclitaxel and Gemcitabine
Number analyzed (Participants) | 40
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 70 [64 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 31
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: defined as the percentage of patients with complete or partial responses based on RECIST 1.1, at any time prior to disease progression, out of all evaluable patients. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Albumin-Bound Paclitaxel and Gemcitabine
Number analyzed (Participants) | 40
Participants
  Partial Response | 18
  Complete Response | 1
  Not Evaluated, withdrew from study | 5
  Stable Disease | 12
  No Response | 4

2. Secondary Outcome: Participants Evaluated for Toxicity
Description: AE's will be collected, tabulated according to CTCAE version 4.0 and summarized using descriptive statistics.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Albumin-Bound Paclitaxel and Gemcitabine
Number analyzed (Participants) | 40
Participants
  Evaluable for toxicity | 37
  Not evaluable for toxicity | 3

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Albumin-Bound Paclitaxel and Gemcitabine
All-Cause Mortality (participants affected / at risk) | 21/40
Serious Adverse Events (participants affected / at risk) | 7/40
Other Adverse Events (participants affected / at risk) | 37/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Albumin-Bound Paclitaxel and Gemcitabine (N=40)
Acute Kidney Injury (Renal and urinary disorders) | 2
Anemia (Blood and lymphatic system disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Creatinine increased (Investigations) | 2
Death NOS (General disorders) | 6
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Edema limbs (General disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Fever (General disorders) | 3
Hip fracture (Injury, poisoning and procedural complications) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypotension (Vascular disorders) | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Infections and infestations - Other, specify (Infections and infestations) | 1
Lung infection (Infections and infestations) | 5
Mucosal Infection (Infections and infestations) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Platelet count decreased (Investigations) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Seizure (Nervous system disorders) | 1
Skin infection (Infections and infestations) | 2
Sudden death NOS (General disorders) | 1
Superficial thrombophlebitis (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Transient ischemic attacks (Nervous system disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Ventricular arrhythmia (Cardiac disorders) | 1
White blood cell decreased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Albumin-Bound Paclitaxel and Gemcitabine (N=40)
Activated partial thromboplastin time prolonged (Investigations) | 5
Alanine aminotransferase increased (Investigations) | 28
Alkaline phosphatase increased (Investigations) | 11
Anemia (Blood and lymphatic system disorders) | 37
Aspartate aminotransferase increased (Investigations) | 25
Blood bilirubin increased (Investigations) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Creatinine increased (Investigations) | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Fatigue (General disorders) | 4
Hypercalcemia (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 37
Hyperkalemia (Metabolism and nutrition disorders) | 12
Hypernatremia (Musculoskeletal and connective tissue disorders) | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 35
Hypocalcemia (Metabolism and nutrition disorders) | 19
Hypoglycemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 9
Hyponatremia (Metabolism and nutrition disorders) | 16
Hypophosphatemia (Metabolism and nutrition disorders) | 2
INR increased (Investigations) | 13
Lymphocyte count decreased (Investigations) | 24
Nausea (Gastrointestinal disorders) | 3
Neutrophil count decreased (Investigations) | 15
Platelet count decreased (Investigations) | 25
White blood cell decreased (Investigations) | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-12): https://cdn.clinicaltrials.gov/large-docs/53/NCT02525653/Prot_SAP_000.pdf